CLINICAL TRIAL: NCT02457117
Title: A Multi-Institutional Registry for CyberKnife Stereotactic Accelerated Partial Breast Irradiation (CK-SAPBI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-0098
Record Dates: First submitted 2015-05-27; First posted 2015-05-29 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Breast Cancer
Keywords: CyberKnife; Partial breast irradiation; accelerated partial breast irradiation; breast sbrt
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: CyberKnife Stereotactic Accelerated Partial Breast Irradiation (CK-SAPBI) — Five fraction radiation therapy to the lumpectomy cavity
  Other Names: Breast SBRT; partial breast irradiation

SUMMARY:
This study is a registry to monitor quality of life and clinical outcomes in patients with clinically localized breast cancer who have received stereotactic accelerated partial breast irradiation via CyberKnife.

DETAILED DESCRIPTION:
Radiotherapy for breast cancer is delivered using several whole breast and partial breast approaches. The optimal approach is unknown. The utilization of partial breast irradiation is growing due to the convenience of fewer fractions versus fifteen- thirty treatments required with conventional or hypofractionated whole breast radiation therapy.

Early results with partial breast techniques are promising, showing similar cancer control and toxicity. There is a large body of mature Phase I/II and preliminary Phase III data available exploring the replacement of WBI with an accelerated course of radiation therapy restricted to the region around the tumor bed (accelerated Partial Breast Irradiation, aPBI) using a variety of techniques. For appropriately selected patients treated with modern techniques, the results are encouraging and the techniques have been shown to be safe, tolerable, and highly reproducible with outcomes similar to WBI.

Currently, there is limited data assessing the quality of life, cosmetic and oncologic outcomes following stereotactic partial breast irradiation in a large patient population. Our study will be the first essential step in aggregating the outcomes of patients undergoing this type of external beam irradiation in a large patient population.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible to participate in the registry if they receive CK-SAPBI in 5 fractions within 12 weeks of surgery and sign an institution specific consent form.

Additionally, subjects will be considered standard risk and optimal for CK-SAPBI if they meet the following criteria:

* Newly diagnosed AJCC (seventh edition) Stage 0 or I breast cancer.
* On histological examination, the tumor must be DCIS or invasive non-lobular carcinoma of the breast
* Surgical treatment of the breast must have been wide excision, lumpectomy or partial mastectomy
* Age 50 years or greater
* ER positive
* PR positive
* Her2 negative (IHC 0-1+; for IHC 2+, FISH must be non-amplified)
* Subjects with invasive tumors should undergo axillary sentinel lymph node evaluation or axillary lymph node dissection.
* Negative inked surgical margins of excision or re-excision, clear of invasive tumor and DCIS by at least 2 mm
* Negative post-excision or post-reexcision mammography if cancer presented with malignancy-associated microcalcifications with no remaining suspicious calcifications in the breast before radiotherapy. Alternatively, a specimen radiograph can be obtained showing all the suspicious calcifications.
* No involved axillary lymph nodes, N0(i+) allowed
* Target lumpectomy cavity/whole breast reference volume must be <30% based on treatment planning CT

Exclusion Criteria:

* -Patients with invasive lobular carcinoma or nonepithelial breast malignancies such as sarcoma or lymphoma.
* Patients with tumors greater than 2 cm
* Patients with surgical margins which cannot be microscopically assessed or not cleared by at least 2mm at pathological evaluation.
* Patients with multicentric carcinoma or with other clinically or radiographically suspicious areas in the ipsilateral breast unless confirmed to be negative for malignancy by biopsy. Breast MRI will be required to exclude multicentric disease and additional suspicious areas will require biopsy to exclude malignancy.
* Patients with involved axillary nodes.
* Patients with collagen vascular diseases (active).
* Patient with known deleterious BRCA1/2 mutations or known mutations in other high penetrance genes (TP53, STK11, PTEN, CDH1)
* Patients with prior ipsilateral breast irradiation.
* Patients with prior ipsilateral thoracic irradiation.
* Patients with Paget's disease of the nipple.
* Patients with diffuse suspicious microcalcifications.
* Patients with suspicious microcalcifications remaining on the post-excision mammogram.
* Patients receiving (neo)adjuvant systemic therapy other than hormonal therapy
* Patients with oncoplastic reconstruction and absence of surgical clips

Ages: 50 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women receiving breast cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
In breast failure | 5 years
  To evaluate the in-breast local failure (Ipsilateral breast events) and patterns of in-breast failure following CK-SAPBI

SECONDARY OUTCOMES:
Cosmesis | 5 years
  Treatment related Cosmesis based on the Harvard Cosmesis Scale
Regional Recurrence | 5 years
  Regional recurrence free interval defined as time from end of radiation treatment to the diagnosis of disease in the regional lymph nodes
Distant Recurrence | 5 years
  Distant disease free interval defined as the time from end of radiation treatment to first diagnosis of distant disease, regardless of the occurrence of any intervening local or regional failure, contralateral breast cancer, or non-breast second primary cancer
Adverse reactions | 5 years
  Toxicity from treatment based on CTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States